CLINICAL TRIAL: NCT03767595
Title: Post Approval Study of the ProACT™ Adjustable Continence Therapy for Men
Brief Title: ProACT Post-Approval Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uromedica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAS001
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ProACT Adjustable Continence Therapy for Men (Experimental): Patients implanted with ProACT Adjustable Continence Therapy for Men
  Interventions: Device: ProACT Adjustable Continence Therapy for Men

INTERVENTIONS:
Device: ProACT Adjustable Continence Therapy for Men — The ProACT therapy consists of two small, adjustable silicone balloons connected with tubing to a port. During a minimally invasive outpatient procedure, the balloons are surgically placed in the area where the prostate was removed or resected.

SUMMARY:
The ProACT Post Approval Study is a 5-year prospective, open-label, multi-center study designed to evaluate the long-term incidence of urethral stricture and device erosion after ProACT implantation. In addition, the study will evaluate whether treatment with ProACT affects clinical outcomes after subsequent SUI therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male of at least 50 years of age.
2. Subject demonstrates stress urinary incontinence.
3. Subject has undergone a radical prostatectomy, transurethral resection of the prostate, or other prostate surgery.
4. Subject is willing and able to undergo surgical implantation of ProACT devices.
5. Subject is willing and able to comply with study-required

   follow-up activities, including annual telephonic follow -up interviews, for a period of 5 years from their date of initial implantation. This includes compliance even after possible explant of ProACT devices and/or possible implantation of subsequent therapies.
6. Subject is willing and able to sign the approved informed consent.
7. Subject has two positive 24-hour pad weight tests (greater than or equal to 8 gram pad weight increase demonstrated in two 24-hour pad weight tests).
8. Subject has a negative urine culture.
9. Subject has no known urogenital malignancy, other than previously treated prostate cancer.
10. Subject meets ONE of the following criteria:

    1. Baseline Prostate-Specific Antigen (PSA) of less than or equal to 2.5ng/mL;
    2. Baseline PSA > 2.5ng/mL and less than or equal to 10 ng/mL AND free PSA greater than or equal to 25% of total PSA;
11. Physician determines subject to be a suitable surgical candidate.

Exclusion Criteria:

1. Subject has an existing urethral stricture, a history of any urethral strictures, or has ever had a urethrotomy.
2. Subject has undergone prostate surgery or any anti-incontinence surgery within the last 12 months.
3. Subject has an artificial urinary sphincter or any components of a previously implanted artificial urinary sphincter in vivo.
4. Subject has undergone radiation therapy in the prostatic area within the last 12 months.
5. Subject has untreated or unsuccessfully treated detrusor instability or over-activity.
6. Subject has an atonic bladder.
7. Subject had, presently has, or is suspected of having bladder cancer.
8. Subject has untreated or unsuccessfully treated bladder stones.
9. Subject has detrusor sphincter dyssynergia.
10. Subject has known hemophilia or a bleeding disorder.
11. Subject has a known severe contrast solution allergy (e.g., anaphylaxis, cardiac, or respiratory arrest).
12. Subject has insulin-dependent diabetes that is uncontrolled or not controllable, as indicated by an A1c test result of = 6.5%.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Urethral Strictures | 5 years
  Cumulative incidence of ProACT-related clinically relevant urethral strictures over 5 years of follow up.
Device Erosions | 5 years
  Cumulative incidence of ProACT device erosions over 5 years of follow-up.
Incontinence Quality of Life Questionnaire (I-QoL) | 5 years
  Results on Validated Incontinence Quality of Life Questionnaire

OTHER OUTCOMES:
Effect of ProACT on Subsequent Stress Urinary Incontinence(SUI) Therapy | 5 years
  This data will be collected with a "Post ProACT Explant Subsequent Therapy Questionnaire".
  This questionnaire will ask 3 questions regarding the ProACT therapy
  1. Did the ProACT therapy have a detrimental effect on the difficulty of the subsequent implant surgery?
  2. Did the ProACT therapy significantly increase the time required to implant the subsequent implant surgery?
  3. Did the ProACT therapy increase the surgical complication rate during the subsequent implant surgery?
  The scale for each question is 0-1. 0 Meaning no effect (a "No" response on the questionnaire) and 1 being some effect ("Yes" response on the questionnaire). No effect (0) on subsequent SUI therapies is the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy C Cook, PhD, Study Director — Uromedica, Inc.
Locations (6):
- United States (6):
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - CentraCare- St. Cloud, Saint Cloud, Minnesota